CLINICAL TRIAL: NCT05507996
Title: An Investigator-initiated Trial Evaluating the Efficacy and Safety of Recombinant Adeno-associated Virus Administration in Patients With Menkes Syndrome
Brief Title: Recombinant Adeno-associated Virus Administration for Patients With Menkes Syndrome
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The PI decides to stop.
Sponsor: Kunming Hope of Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE-1
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Menkes Syndrome
Keywords: gene therpy; adeno-associated virus
MeSH Terms: conditions — Menkes Kinky Hair Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-arm study of recombinant adeno-associated virus (Experimental): An open, single-arm study of recombinant adeno-associated virus
  Interventions: Drug: Recombinant adeno-associated virus administration

INTERVENTIONS:
Drug: Recombinant adeno-associated virus administration — The investigational medical product will be injected from 1E12 GC/kg to 1E14 GC/kg.

SUMMARY:
It is a single-center, open, single-arm, non-randomized investigator-initiated trial evaluating the efficacy and safety of recombinant adeno-associated virus administration for patients with Menkes syndrome.

DETAILED DESCRIPTION:
Who can participate? Patients with Menkes syndrome were diagnosed by combining clinical and genetic diagnoses.

How to conduct this study? In this study, the constructed recombinant adeno-associated virus preparation will be delivered to patients with Menkes syndrome. After administration, close follow-up will be conducted for at least three months, followed by regular follow-up until at least the 12th month. The efficacy and safety of treatment will be observed and evaluated. After the completion of the study, participants will decide whether to participate in the long-term follow-up program for five years.

What are the possible benefits and risks of participating? Benefits: This study may prolong the life span and improve the prognosis of Menkes syndrome subjects. The information obtained from this study will help determine what treatment may be safe and effective for other subjects with similar conditions.

Risks: Subjects may have adverse reactions to the treatment. These adverse reactions may include abnormal liver injury, fever, thrombocytopenia, thrombotic microangiopathy, and possibly others.

Where is the study run? Kunming Hope of Health Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. The definitive diagnosis of Menkes disease is determined by molecular genetic confirmation of ATP7A mutations.
2. Disorder of copper metabolism with the serum copper < 50 ug/dl (reference 70-180 ug/dl) and ceruloplasmin < 20 mg/dl (reference 20-45 mg/dl) in the absence of copper supplement injection.
3. Clinical onsets of developmental retardation, seizures, and hypotonia with delay in poor head control and inability to sit at the age of 2-3 months.
4. willingness to complete the informed consent process and to comply with study procedures and visit schedule.
5. willingness to agree with the demand of nasal or gastrostomy feeding for nutrition maintenance in the opinion of the investigator.

Exclusion Criteria:

1. Inability to be accepted for delivering the Investigational medical product due to failure to recover from severe or acute diseases.
2. Presence of specific anti-AAV antibodies.
3. Active viral infection (includes HIV, COVID-19, or serology positive for hepatitis B or C).
4. Allergy to the substance or excipients in the Investigational medical product solution.
5. Previous or current participation in any other gene therapies.
6. Severe abnormality of hepatic, renal, and cardiac function.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Monitoring the disease course or vital signs to assess the efficacy of the investigational medical product | Up to the end of life after infusion or 12 months after the age of 3 years
  Based on studies of the natural history of Menkes syndrome, which shows that patients have a life span of fewer than three years, this study will evaluate the endpoint of life of patients with the investigational medical product infusion. The endpoint of life is defined as death or the need for ventilatory support (device dependence of at least 16 hours per day for more than 14 days).
Incidence of adverse events(AE) after the investigational medical product infusion | Up to 12 months after the investigational medical product infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included. Description, time, classification, and outcome of AE events resulted from the investigational medical product, delivery method, or emergency measures will be recorded in the case report form.

SECONDARY OUTCOMES:
Developmental behavior assessment | At baseline and 3, 6, 9, 12 months after infusion
  CHOP INTEND was developed to be used on children from 3 months to over four years, although it is not limited to this age range. It was developed by looking at babies with SMA Type 1 and infants with other similar conditions, such as Menkes syndrome. There are 16 parts, and the scale scores infants on how well they can perform certain movements or what the physiotherapist sees while watching the child. Each one is scored from 0 to 4, with 0 being no response/ability to perform the movement and 4 being 'complete response' (being able to perform the task). The total possible score is 64.
  The Developmental Behavior Scale for Children aged 0-6 years (WS/T 580-2017) released by the Ministry of Health of China is used to monitor and evaluate the development improvement of patients in gross motor, fine motor, language, adaptive ability, and social behavior. The scale applies to children aged 0-6 years, with 8-10 test items in each group, totaling 261.
Weight | At baseline and 3, 6, 9, 12 months after infusion
  Record weight of patients in kilograms
Height | At baseline and 3, 6, 9, 12 months after infusion
  Record height of patients in meters
Head circumference | At baseline and 3, 6, 9, 12 months after infusion
  Record head circumference of patients in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, Principal Investigator — Kunming Hope of Health Hospital
Locations (1):
- Kunming Hope of Health Hospital, Kunming, Yunnan, China